CLINICAL TRIAL: NCT03248102
Title: Finding Evidence to Treat Or Reassure in Appendicitis (FETOR)
Acronym: FETOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PS15/261
Record Dates: First submitted 2017-07-04; First posted 2017-08-14 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Appendicitis
Keywords: paediatric
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with suspected appendicitis (Experimental): Patients with suspected appendicitis Aged 5 and up to their 16th birthday on arrival to A&E
  Interventions: Diagnostic Test: Blowing into the mouthpiece

INTERVENTIONS:
Diagnostic Test: Blowing into the mouthpiece — Blowing into the mouthpiece of diagnostic device

SUMMARY:
Acute appendicitis is the most common surgical emergency in childhood. Despite access to current diagnostic modalities, diagnosis may be challenging since the child may have difficulty in articulating symptoms. Additionally there is a high frequency of atypical presentation and rapid progression. Delayed diagnosis in children is reported as being up to 60%. Delayed diagnosis >48hr increases the perforation rate from 21% to 71%. Around 20% of children presenting with appendicitis have perforated by the time they come to surgery.

Appendix perforation is associated with a prolonged hospital stay and increased cost. Once perforated, major complication rates increase from 1.2% to 6.4%, median bed stay increases from 2 to 6 days and hospitalisation costs are estimated at US $33,348.

Conversely, a false positive diagnosis leads to unnecessary surgery in 12%. It has been suggested that only 35% of surgical referrals with possible appendicitis actually need surgery thus impacting on resource use.

A reliable test, especially if painless, would be very useful. If positive the child could undergo early appendicectomy in expectation of a reduction in the perforation rate (and, therefore, reduction in hospital stay). If negative the child could be discharged home safely. No adequate biomarker has been identified.

Technology already exists to detect changes in Volatile Organic Compounds (VOC) in gases. VOC analysis is already used commercially to identify disease processes in animals and crops. Although VOC has been previously used to detect human diseases, it has never been used to look for changes in the composition of breath in appendicitis.

The investigators hypothesise that the composition of VOC's in children with appendicitis will differ from those without. The investigators anticipate these differences will be of diagnostic and prognostic value in clinical practice. The feasibility of collecting breath samples from children with possible appendicitis to allow VOC testing has not been examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected appendicitis
* Aged 5 and up to their 16th birthday on arrival to A&E
* Patients referred to the Paediatric surgical team that have presented to the Leeds General Infirmary through A&E, the Children's Assessment Unit, or via direct referral from another team or hospital.
* Consecutive presentations who can have some or all of VOC sampling during working week.

Exclusion Criteria:

* Patients with known alternative cause of abdominal pain (e.g. known Inflammatory Bowel Disease)
* Patients who are both admitted and discharged when no researcher is available

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Breath collection for analysis | 3 minutes
  Collect breath from children with abdominal pain meeting inclusion criteria assess ment to changes in Volatile Organic Compounds (VOC)

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom

REFERENCES:
- [Derived] Wong DC, Relton SD, Lane V, Ismail M, Goss V, Bytheway J, West RM, Deuchars J, Sutcliffe J. Bedside breath tests in children with abdominal pain: a prospective pilot feasibility study. Pilot Feasibility Stud. 2019 Nov 5;5:121. doi: 10.1186/s40814-019-0502-x. eCollection 2019. PMID 31720000